CLINICAL TRIAL: NCT05641987
Title: CPH-NEW IV - Total Worker Health - Total Teacher Health
Brief Title: Effectiveness of the Educator Well-being Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer Cavallari, Associate Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-123S-2; 1 U19OH012299-01-00 (Other Grant/Funding Number: National Institute for Occupational Safety and Health); 1U19OH012299-01 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Participatory Action Research; Occupational Health; Educator Well-being; Employee Health

STUDY DESIGN:
Intervention Model Description: A stepped wedge design (prospective cohort with concurrent controls) among six paired, elementary schools, implement and evaluate the Total Teacher Health Toolkit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educator Well-being Program (Experimental): Staff at participating schools will experience the Educator Well-being Program process and complete pre- and post-intervention survey.
  Interventions: Behavioral: Healthy Workplace Participatory Program
- Delayed Intervention (Active Comparator): Status quo program remains in place with new ongoing data collection, then experimental intervention as above.
  Interventions: Behavioral: Healthy Workplace Participatory Program

INTERVENTIONS:
Behavioral: Healthy Workplace Participatory Program — The Center for the Promotion of Health in the New England Workplace's (CPH-NEW's) Healthy Workplace Participatory Program (HWPP) is a participatory process in which end-users design TWH interventions that simultaneously change organizational and individual behavior to improve the health, safety and well-being of their workforce. The HWPP uses a process to empower workers to identify the root causes of health and safety concerns and then design, implement and evaluate interventions to address those problems. The Total Teacher Health Project adapted the HWPP for educators and refer to it as the Educator Well-being Program.

SUMMARY:
Using a stepped wedge design (prospective cohort with concurrent controls) among six paired, elementary schools, investigators will implement and evaluate the Educator Well-being Program. The investigators will evaluate whether the process improves organizational-level factors, teacher mental well-being (stress, depression and anxiety symptoms).

ELIGIBILITY:
Inclusion Criteria:

* All staff aged 18 years or older at the time of survey administration within the three school districts will be eligible for participation.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Work Stress | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey for Educators" includes 1 question related to stress (Eddy, 2009). The score ranges from 1-10, where higher scores indicate more stress.
Perceived Stress | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey for Educators" includes 10 items from the Perceived Stress Scale (Cohen, 1983). A summary score is created with score ranges from 0-40, where higher scores indicate more stress.
Anxiety Symptoms | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey for Educators" includes 7 items from the GAD-7 (Spitzer et al., 2006). A summary score is created and scores range from 0-21, where higher scores indicate greater anxiety symptoms.
Depression Symptoms | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey Educator" includes 10 from the CES-D (Radloff et al., 1977) A summary score is created by summing items score ranges from 0-30, where higher scores indicate greater depression symptoms.
Well-being | Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 2 items adapted from the SF-36. One item assesses physical health, the other mental health with both on a scale from 1 (poor) to 5 (excellent) A summary score is created by averaging the two items with a range from 1-5, where higher scores indicate better well-being.
Burnout (Emotional Exhaustion) | Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 9 items from Maslach Burnout Inventory for Educators (Maslach 1996). A summary score is created by summing the nine items, after reverse coding as required, with a range from 0-54, where higher scores indicate higher burnout.
Burnout (Personal Accomplishment) | Frame: Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 8 items from Maslach Burnout Inventory for Educators (Maslach 1996). A summary score is created by summing the nine items, after reverse coding as required, with a range from 0-48, where lower scores indicate higher burnout.
Burnout (Depersonalization) | Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 5 items from Maslach Burnout Inventory for Educators (Maslach 1996). A summary score is created by summing the nine items, after reverse coding as required, with a range from 0-30, where higher scores indicate higher burnout.
Work-life conflict | Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 1 item on work-life conflict (Waumsley, 2010). The item is assessed on a scale from 1 to 5 (strongly disagree to strongly agree) where higher scores indicate higher work-life conflict.
Intention to Turnover | Prior to random selection of immediate and delayed intervention site, and 1 year later
  The "All-Employee Survey for Educators" includes 2 items to assess turnover intention (Hurrell, 1998). The items are assessed on a scale from 1 to 5 (strongly disagree to strongly agree) and averaged where higher scores indicate higher intent to turnover.

SECONDARY OUTCOMES:
Change in Team Attendance | Through study completion, an average of two years
  Attendance for each Educator Design Team meeting (1-4 times per month)
Change in Team Engagement | Through study completion, an average of two years
  Percentage of combined agree and strongly agree responses for 1 survey item collected following Educator Design Team meetings (1-4 times per month): "The discussion was meaningful for achieving health, safety, and well-being goals." (Strongly Agree, Agree, Disagree, Strongly Disagree, Not Applicable). Items are computed individually.
Change in Level of Committee Activity | Through study completion, an average of two years
  A qualitative summary of field notes collected by research personnel following Educator Design Team and Administrator Team meetings (1-4 times per month) over the course of the study.
Change in team-selected health/safety/well-being issue | Through study completion, an average of two years
  Targeted pre- and post-intervention surveys will be designed and administered by the Educator Design Team
Proportion of content followed according to the Educator Well-being Program protocol | Through study completion, an average of two years
  A process measure that will be determined by adherence to Educator Well-being Program protocol and pre-designed agendas for Educator Design Team meetings (1-4 times per month)
Supportive health climate | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey Educator" includes 3 items from Multi-faceted organizational health climate assessment (Zweber et al., 2018). A summary score is created by averaging the 3 items with score ranges from 1-4, where higher scores indicate more supportive health climate.
Supportive School Climate | Prior to random selection of immediate and delayed intervention site, and 1 years later
  The "All-Employee Survey Educator" includes 6 from the School Climate sub-scale for staff connection (La Salle et al. 2018) A summary score is created by averaging the items with score ranges from 1-4, where higher scores indicate a greater more supportive school climate.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cavallari, ScD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No